CLINICAL TRIAL: NCT06277986
Title: Clinical Value of Tumor Cell-derived Exosomal miRNA in Early Diagnosis of Gastric Cancer Cachexia
Brief Title: Early Diagnosis of Gastric Cancer Cachexia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212018-F-2
Record Dates: First submitted 2022-01-16; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia | interventions — dermcidin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer patients with non-cachexia
  Interventions: Other: cachexia
- Gastric cancer patients with cachexia
  Interventions: Other: cachexia

INTERVENTIONS:
Other: cachexia — Cachexia mainly manifests as weight loss. 1)weight loss >5% over past 6 months. 2)BMI<20 and any degree of weight loss >2%. 3)Appendicular skeletal muscle index consistent with sarcopenia and any degree of weight loss >2%.

SUMMARY:
Gastric cancer is one of the most common malignancies, the morbidity and mortality of which are among the highest. In cancer patients, the incidence of cachexia is very high, and even 80% of patients will eventually develop into cachexia. However, once gastric cancer patients develop cachexia, patients are unlikely to obtain clinically significant benefits from conventional treatment. Therefore, it is important to find biomarkers for early detection of cachexia. The investigators carried out a plasma-derived exosomal microRNA(miRNA) study for early diagnosis of cachexia in gastric cancer, and the development of early diagnosis kits for gastric cancer cachexia.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies, the morbidity and mortality of which are among the highest. In gastric cancer patients, the incidence of cachexia is very high, and even 80% of patients will eventually develop into cachexia. However, once gastric cancer patients develop cachexia, patients are unlikely to obtain clinically significant benefits from conventional treatment. Therefore, it is important to find biomarkers for early detection of cachexia. The investigators carried out a plasma-derived exosomal microRNA(miRNA) study for early diagnosis of cachexia in gastric cancer, and the development of early diagnosis kits for gastric cancer cachexia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gastric cancer diagnosed by histopathology or cytopathology
2. Complete clinical and pathological data
3. No previous or current mental illness or disturbance of consciousness

Exclusion Criteria:

1. With multiple tumors or other malignant diseases
2. Combined with other chronic wasting and metabolic diseases
3. Past patients with non-tumor cachexia
4. People with mental illness or unable to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research object is patients with confirmed gastric cancer.According to diagnostic criteria, patients are divided into cachexia group and non-cachexia group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
BMI | six months
  Calculate BMI based on changes in body weight in the past six months

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China